CLINICAL TRIAL: NCT01586650
Title: Effects of Aerobic Training in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Martin F Simoes, MD, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1325/08
Record Dates: First submitted 2012-04-21; First posted 2012-04-27 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Ankylosing Spondylitis
Keywords: ankylosing spondylitis; aerobic exercise
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic training (Experimental): The patients in this arm perform a 50-minute-walking at anaerobic threshold plus stretching exercises 3 times a week for 12 weeks.
  Interventions: Other: aerobic training; Other: Stretching exercises
- Stretching exercises (Placebo Comparator): The control group perform global stretching exercises for approximately 20 minutes 3 times a week for 12 weeks.
  Interventions: Other: Stretching exercises

INTERVENTIONS:
Other: aerobic training — The intervention comprises fifty minutes of walking at anaerobic threshold plus stretching exercises 3 times a week for 12 weeks.
  Arms: Aerobic training
Other: Stretching exercises — Global stretching exercises will be performed for about 20 minutes 3 times a week for 12 weeks with supervision of specialized physiotherapists.

SUMMARY:
This is a randomized controlled trial with blinded assessor on the effects of aerobic exercise (walking)in patients with Ankylosing Spondylitis.

DETAILED DESCRIPTION:
Ankylosing Spondylitis (AS) is a systemic inflammatory disease that affects mainly the spine and compromises globally the physical capacity of the patients. Despite new advances in pharmacological therapy, physiotherapy and exercise remain essential in the treatment of AS. However, the literature lacks studies showing which types of exercises are more effective in patients with AS.

This is a randomized controlled trial with the objective is to evaluate the effects of aerobic training on functional capacity, mobility, disease activity, cardiopulmonary capacity and cytokine levels (TNF, IL10, IL6 and IL1) in patients with AS.

The duration of the trial is 24 weeks with the first 12 weeks reserved to exercise programs. The participants will be divided in two groups. The intervention group (IG) will perform walking for 50 minutes plus global stretching 3 times a week for 12 weeks. The control group (CG) will do only stretching exercises 3 times a week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ankylosing Spondylitis according to New York modified criteria.

  * Stable drug treatment for at least 3 months
  * Sedentary for at least 3 months before randomization
  * Steinbrocker class I/II

Exclusion Criteria:

* Uncontrolled Systemic Arterial Hypertension and Diabetes mellitus.

  * Ischemic heart disease
  * Clinically significant diseases
  * Orthopedic surgery, such as hip arthroplasty, in the last year.
  * Inability to walk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in BASFI | Baseline, after 6, 12 and 24 weeks.
  Bath Ankylosing Spondylitis Functional Index (BASFI) is a quaestionnaire with 10 questions about functional capacity validated to AS patients. Each question is answered with a visual analogue scale 0-10 cm. Zero means the best, and 10 the worst function.

SECONDARY OUTCOMES:
Change in BASDAI | Baseline, after 6, 12 and 24 weeks.
  Bath Ankylosing Spondylitis Disease Activity Score (BASDAI) is a instrument with 6 questions about disease activity validated to AS patients. The questions comprise the following areas: back pain, peripheral pain, morning stifness, fatigue and enthesitis.
Change in BASMI | Baseline, after 6, 12 and 24 weeks.
  Bath Ankylosing Spondylitis Mobility Index (BASMI) is an instrument that comprises 5 measures of mobility validated to AS patients. The measurements are: cervical rotation, lumbar flexion (Schober's test modified, intermalleolar distance, lumbar side flexion and tragus to wall. The total score is shown in a 0-10 cm visual analogue scale. The low scores represent better mobility.
Change in HAQ-S | Baseline, after 6, 12 and 24 weeks.
  Health Assessment Questionnaire for Spondyloarthritis (HAQ-S)is a questionnaire with 10 domains about functional capacity validated to AS patients. The scores ranges from 0 to 3.
Incremental cardiopulmonary exercise testing protocol by treadmill | Baseline and after 12 weeks.
  Incremental cardiopulmonary exercise testing protocol by treadmill is used to measure aerobic capacity of the patients.
Levels of C reactive protein and erythrocyte rate sedimentation | Baseline, after 6. 12 and 24 weeks
  CRP and ESR are laboratory methods to evaluate inflammatory response using blood sample.
Levels of cytokines- TNF, IL10, IL6 and IL1. | Baseline and after 12 weeks.
  Cytokines are substances that make part of inflammatory response. The most important cytokines- TNF alpha, IL10, IL6 and IL1 will be measured in serum samples.
Change in the Six minute walking test | Baseline, after 6, 12 and 24 weeks.
  The 6-minute walking test is a instrument to evaluate functional capacity. It is performed measuring the distance that the participant is able to walk during 6 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Natour, Prof, MD, Study Director — Federal University of São Paulo
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Braun J, van den Berg R, Baraliakos X, Boehm H, Burgos-Vargas R, Collantes-Estevez E, Dagfinrud H, Dijkmans B, Dougados M, Emery P, Geher P, Hammoudeh M, Inman RD, Jongkees M, Khan MA, Kiltz U, Kvien T, Leirisalo-Repo M, Maksymowych WP, Olivieri I, Pavelka K, Sieper J, Stanislawska-Biernat E, Wendling D, Ozgocmen S, van Drogen C, van Royen B, van der Heijde D. 2010 update of the ASAS/EULAR recommendations for the management of ankylosing spondylitis. Ann Rheum Dis. 2011 Jun;70(6):896-904. doi: 10.1136/ard.2011.151027. PMID 21540199